CLINICAL TRIAL: NCT01421186
Title: A Phase 1/2a, Open-Label, Multicentre, Dose-Escalation Study to Evaluate the Safety and Preliminary Efficacy of the Human Anti-CD 38 Antibody MOR03087 as Monotherapy and in Combination With Standard Therapy in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: A Phase 1/2a Study of Human Anti-CD 38 Antibody MOR03087 (MOR202) in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR202C101; DRKS00003145 (Registry Identifier: German Clinical Trail Register)
Record Dates: First submitted 2011-07-29; First posted 2011-08-22 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; MOR03087 (MOR202); Lenalidomide; Pomalidomide; CD38
MeSH Terms: conditions — Multiple Myeloma | interventions — felzartamab; Dexamethasone; pomalidomide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 dose escalation (Experimental): Part A: MOR03087 dose escalation; biweekly treatment
  Part B: MOR03087 dose escalation; weekly treatment
  Part C: MOR03087 dose escalation (weekly treatment) + dexamethasone
  Part D: MOR03087 weekly treatment in combination with pomalidomide + dexamethasone
  Part E: MOR03087 weekly treatment in combination with lenalidomide + dexamethasone
  For all parts, patients will be treated until disease progression (PD) or until a maximum of 3 years after first treatment.
  Interventions: Drug: MOR03087 phase 1 dose escalation; Drug: Dexamethasone; Drug: Pomalidomide; Drug: Lenalidomide
- Phase 2a confirmatory cohorts (Experimental): Confirmatory cohorts of MOR03087 monotherapy (plus or minus dexamethasone), in combination with pomalidomide plus dexamethasone, and in combination with lenalidomide plus dexamethasone.
  Following completion of Parts A, B, and C (dose escalation of MOR03087 biweekly and weekly schedules), the Maximum Tolerated Dose (MTD) or recommended dose and dosing regimen will be confirmed in a minimum of 6 subjects.
  Following completion of Parts D (dose escalation of MOR03087 in combination with pomalidomide + dexamethasone) and E (dose escalation of MOR03087 in combination with lenalidomide + dexamethasone), the MTD and/or recommended dose in each part will be confirmed in a minimum of 6 subjects.
  For all parts, patients will be treated until PD or until a maximum of 3 years after first treatment.
  Interventions: Drug: MOR03087; Drug: Dexamethasone; Drug: Pomalidomide; Drug: Lenalidomide

INTERVENTIONS:
Drug: MOR03087 phase 1 dose escalation — Treatment cycles will be 28 days. Initial MOR03087 doses will be 0.01 mg/kg in part A, 4 mg/kg in parts B and C and 8 mg/kg in parts D and E; in all parts MOR03087 doses will be escalated to a maximum of 16 mg/kg. In part A, patients will receive a biweekly intravenous infusion of MOR03087 which will be administered on days 1 and 15 of the cycle. In parts B to E patients will receive a weekly intravenous infusion of MOR03087 which will be administered on days 1, 8, 15, and 22 of the cycle.
  In all parts a loading dose of MOR03087 will be additionally administered on day 4 of cycle 1.
  Arms: Phase 1 dose escalation
Drug: MOR03087 — MOR03087 will be administered according to the Maximum Tolerated Dose (MTD) or recommended dose and dosing regimen for MOR03087 from parts A-E of the phase I dose escalation. The biweekly MOR03087 regimen as described in part A; the weekly regimen as described for parts B-E.
  Arms: Phase 2a confirmatory cohorts
Drug: Dexamethasone — Dexamethasone will be administered to patients orally; 40 mg (≤ 75 years old) or 20 mg (> 75 years old) on days 1, 8, 15, and 22 of the 28-day cycle. An additional dose will be administered in cycle 1 on day 4.
Drug: Pomalidomide — Pomalidomide will be administered to patients orally 4 mg on days 1-21 of the 28-day cycle.
Drug: Lenalidomide — Lenalidomide will be administered to patients orally 25 mg on days 1-21 of the 28-day cycle.

SUMMARY:
This is an open-label, multicentre, dose escalation study to characterize the safety and preliminary efficacy of the human anti-CD38 antibody MOR03087 (MOR202), in adult subjects with relapsed/refractory multiple myeloma, as monotherapy and in adult subjects with relapsed/refractory multiple myeloma in combination with standard therapy.

DETAILED DESCRIPTION:
The study enrolled patients aged 18 years or older with relapsed or refractory multiple myeloma and Karnofsky performance status of 60% or higher. Patients were assigned to the different treatment regimens with MOR202 ranging between 0·01 mg/kg and 16 mg/kg in a 3 + 3 design. Dose-escalation and expansion was done either with MOR202 intravenous infusions alone (MOR202 q2w [twice a week] and q1w [weekly] groups) or in combination with dexamethasone (MOR202 with dexamethasone group), with dexamethasone plus pomalidomide (MOR202 with dexamethasone plus pomalidomide group) or plus lenalidomide (MOR202 with dexamethasone plus lenalidomide group). Primary endpoints were safety, MOR202 maximum tolerated dose (or recommended dose) and regimen, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years and older
2. Relapsed or refractory multiple myeloma defined as:

   Parts A, B and C:

   (i) Failure of at least 2 previous therapies which must have included an immunomodulatory agent and a proteasome inhibitor (either together or part of different therapies) (ii) All subjects must have documented progression during or after their last prior therapy for multiple myeloma

   Part D:

   (i) At least 2 previous therapies including lenalidomide and a proteasome inhibitor (ii) All subjects must have documented progression during or within 60 days after their last prior therapy for multiple myeloma

   Part E:

   (i) Received at least one previous therapy (ii) All subjects must have documented progression during or after their last prior therapy for multiple myeloma
3. Presence of serum M-protein ≥ 0.5 g per 100 mL (≥ 5 g/L) and / or urine M-protein ≥ 200 mg per 24-hour period
4. Absolute neutrophil count (ANC) ≥ 1,000 / mm3
5. Haemoglobin ≥ 8 g/dL
6. Ability to comply with all study related procedures, medication use and evaluations

Exclusion Criteria:

1. Primary refractory multiple myeloma
2. History of significant cerebrovascular disease or sensory or motor neuropathy of toxicity grade 3 or higher
3. Treatment with systemic investigational agent within 28 days prior to first study treatment
4. Solitary plasmacytoma or plasma cell leukaemia
5. Previous allogenic stem cell transplant (SCT)
6. Prior therapy with other monoclonal antibodies targeting the CD38 antigen or prior therapy with other IgG monoclonal antibodies within 3 months prior to first study treatment, or IgM monoclonal antibodies within 1 month prior to first study treatment
7. Active systemic infection
8. Systemic disease preventing study treatment
9. Multiple myeloma with central nervous system (CNS) involvement
10. Previous treatment with cytotoxic chemotherapy or large field radiotherapy or other myeloma specific therapy within 28 days prior to first study treatment (radiation to a single site as concurrent therapy is allowed)
11. Significant uncontrolled cardiovascular disease or cardiac insufficiency (New York Heart Association [NYHA] classes III, IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- AKH (Allgemeines Krankenhaus der Stadt Wien), Abteilung für Klinische Onkologie, Universitätsklinik für Innere Medizin I, Vienna, Austria
- Germany (9):
  - Charité - Universitätsmedizin Berlin, CBF: Campus Benjamin Franklin, CC 14: Tumormedizin, Medizinische Klinik mit Schwerpunkt Hämatologie, Onkologie, Berlin
  - Medizinische Klinik und Poliklinik I, Universitätsklinikum Carl Gustav Carus, Dresden
  - Medizinische Klinik 5 - Hämatologie und Internist. Onkologie, Universitätsklinikum Erlangen, Erlangen
  - Medizinische Universitätsklinik, Abt. Innere Medizin I, Freiburg im Breisgau
  - Universitäsklinikum Heidelberg, Klin.-Pharmakologisches Studienzentrum, Heidelberg
  - Sektion für Stammzell- und Immuntherapie, II. Medizinischen Klinik,, Kiel
  - Klinikum rechts der Isar/ Studien / III. Med. Klinik, Munich
  - Medizinische Klinik II, Abt. Hämatologie, Onkologie,, Tübingen
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik II, Studienambulanz für Hämatologie/Onkologie und Infektiologie, Würzburg

REFERENCES:
- [Derived] Raab MS, Engelhardt M, Blank A, Goldschmidt H, Agis H, Blau IW, Einsele H, Ferstl B, Schub N, Rollig C, Weisel K, Winderlich M, Griese J, Hartle S, Weirather J, Jarutat T, Peschel C, Chatterjee M. MOR202, a novel anti-CD38 monoclonal antibody, in patients with relapsed or refractory multiple myeloma: a first-in-human, multicentre, phase 1-2a trial. Lancet Haematol. 2020 May;7(5):e381-e394. doi: 10.1016/S2352-3026(19)30249-2. Epub 2020 Mar 11. PMID 32171061

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: MOR03087 Biweekly Dose Escalation: Treatment cycle 28 days, MOR03087 doses applied day 1 & 15, initial 0.01 mg/kg, max 16 mg/kg
- Part B: MOR03087 Weekly Dose Escalation: Treatment cycle 28 days, MOR03087 doses applied day 1, 8, 15 & 22 plus extra dose on day 4 of cycle 1, Initial MOR03087 dose 4 mg/kg, max 16 mg/kg
- Part C: MOR03087 Plus Dexamethasone: Treatment cycle 28 days, iv MOR03087 and oral dexamethasone (DEX) applied day 1, 8, 15 & 22 plus extra dose on day 4 of cycle 1, initial MOR03087 dose 4 mg/kg, max 16 mg/kg. DEX dose 40 mg (≤ 75 years old) or 20 mg (> 75 years old)
- Part D: MOR03087 Plus Pomalidomide + Dexamethasone: Treatment cycle 28 days, iv MOR03087 and oral dexamethasone (DEX) applied day 1, 8, 15 & 22 plus extra dose on day 4 of cycle 1, initial MOR03087 dose 4 mg/kg, max 16 mg/kg. DEX dose 40 mg (≤ 75 years old) or 20 mg (> 75 years old). Pomalidomide was administered to patients orally 4 mg on days 1-21 of the 28-day cycle.
- Part E: MOR03087 Plus Lenalidomide + Dexamethasone: Treatment cycle 28 days, iv MOR03087 and oral dexamethasone (DEX) applied day 1, 8, 15 & 22 plus extra dose on day 4 of cycle 1, initial MOR03087 dose 4 mg/kg, max 16 mg/kg. DEX dose 40 mg (≤ 75 years old) or 20 mg (> 75 years old).
  Lenalidomide was administered to patients orally 25 mg on days 1-21 of the 28-day cycle.
Period: Overall Study
Arm/Group | Part A: MOR03087 Biweekly Dose Escalation | Part B: MOR03087 Weekly Dose Escalation | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone
Started | 31 | 4 | 18 | 21 | 17
Completed | 31 | 4 | 18 | 21 | 17
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part D: MOR03087 Plus Pomalidomide + Dexamethasone: Treatment cycle 28 days, iv MOR03087 and oral dexamethasone (DEX) applied day 1, 8, 15 & 22 plus extra dose on day 4 of cycle 1, initial MOR03087 dose 8 mg/kg, max 16 mg/kg. DEX dose 40 mg (≤ 75 years old) or 20 mg (> 75 years old). Pomalidomide was administered to patients orally 4 mg on days 1-21 of the 28-day cycle.
- Part E: MOR03087 Plus Lenalidomide + Dexamethasone: Treatment cycle 28 days, iv MOR03087 and oral dexamethasone (DEX) applied day 1, 8, 15 & 22 plus extra dose on day 4 of cycle 1, initial MOR03087 dose 8 mg/kg, max 16 mg/kg. DEX dose 40 mg (≤ 75 years old) or 20 mg (> 75 years old).
  Lenalidomide was administered to patients orally 25 mg on days 1-21 of the 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Part A: MOR03087 Biweekly Dose Escalation | Part B: MOR03087 Weekly Dose Escalation | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone | Total
Number analyzed (Participants) | 31 | 4 | 18 | 21 | 17 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 1 | 7 | 10 | 8 | 34
  >=65 years | 23 | 3 | 11 | 11 | 9 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 0 | 8 | 8 | 5 | 33
  Male | 19 | 4 | 10 | 13 | 12 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 31 | 4 | 18 | 21 | 17 | 91
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 0 | 3 | 1 | 0 | 4
  Germany | 31 | 4 | 15 | 20 | 17 | 87

OUTCOME MEASURES:

1. Primary Outcome: Determination of Maximum Tolerated Dose and / or Recommended Dose and Dosing Regimen of MOR03087
Description: 1. as monotherapy
  2. in combination with dexamethasone
  3. in combination with pomalidomide + dexamethasone
  4. in combination with lenalidomide + dexamethasone
Time Frame: First cycle of treatment
Measure: Number; unit: mg/kg
Arm/Group | Part A: MOR03087 Biweekly Dose Escalation | Part B: MOR03087 Weekly Dose Escalation | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone
Number analyzed (Participants) | 31 | 4 | 18 | 21 | 17
mg/kg | 16 | 16 | 16 | 16 | 16

2. Primary Outcome: Number of Participants Who Develop Anti-MOR03087 Antibodies
Description: Number of participants who develop anti-MOR03087 antibodies, a measure of immunogenicity
Time Frame: during treatment period, maximum 3 years after 1st dose
Population: all patients with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MOR03087 Biweekly Dose Escalation | Part B: MOR03087 Weekly Dose Escalation | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone
Number analyzed (Participants) | 31 | 4 | 18 | 21 | 17
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Overall Response Rate
Description: number (#) of patients responding (# stringent complete response + # complete response + # very good partial response + # partial response)
Time Frame: maximum 3 years after 1st dose
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MOR03087 Biweekly Dose Escalation | Part B: MOR03087 Weekly Dose Escalation | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone
Number analyzed (Participants) | 31 | 4 | 18 | 21 | 17
Participants | 0 | 0 | 5 | 10 | 11

4. Secondary Outcome: Time to Progression
Description: Time to Progression (Kaplan Meier estimate)
Time Frame: patients were observed for up to 36 months
Population: safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: MOR03087 Biweekly Dose Escalation | Part B: MOR03087 Weekly Dose Escalation | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone
Number analyzed (Participants) | 31 | 4 | 18 | 21 | 17
months | 1.1 [1.0 to 1.4] | 2.1 [0.7 to NA] — Upper confidence limit could not be estimated due to low number of patients with an event. | 8.4 [1.4 to 11.1] | 15.9 [4.1 to 25.8] | 33.2 [5.1 to NA] — Upper confidence limit could not be estimated due to low number of patients with an event.

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (Kaplan Meier estimates)
Time Frame: patients were observed up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: MOR03087 Biweekly Dose Escalation | Part B: MOR03087 Weekly Dose Escalation | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone
Number analyzed (Participants) | 31 | 4 | 18 | 21 | 17
months | 1.1 [1.0 to 1.4] | 2.1 [0.7 to NA] — Upper confidence limit could not be estimated due to low number of patients with an event. | 8.4 [1.4 to 11.1] | 15.9 [3.0 to 22.1] | 26.7 [5.1 to NA] — Upper confidence limit could not be estimated due to low number of patients with an event.

6. Secondary Outcome: Duration of Response
Description: Duration of response (Kaplan Meier estimates)
Time Frame: patients were observed up to 36 months
Population: Of the total 91 patients, 26 obtained a response: 5 in part C, 10 in part D and 11 in part E. Duration of response was calculated only in these patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone
Number analyzed (Participants) | 5 | 10 | 11
months | 16.7 [1.9 to NA] — Upper confidence limit could not be estimated due to low number of patients with an event. | 21.2 [9.2 to NA] — Upper confidence limit could not be estimated due to low number of patients with an event. | 32.2 [4.2 to NA] — Upper confidence limit could not be estimated due to low number of patients with an event.

7. Secondary Outcome: Pharmacokinetics: Cmax - Maximum Observed Serum Concentration for MOR202
Description: PK analysis for MOR202 4, 8 and 16 mg/kg IV once weekly dose groups only, since serum concentrations of MOR202 were substantially affected by target mediated drug disposition effects for remaining dose groups
Time Frame: up to 7 days after last MOR202 dose
Population: Pharmakokinetics was analysed on all available data on patients receiving 4mg/kg weekly, 8mg/kg weekly and 16 mg/kg weekly irrespective in which part the patients were treated.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- 4 mg/kg QW: Dosing at 4 mg/kg IV once weekly (incl. one add. dose on Cycle 1 Day 4)
- 8 mg/kg QW: Dosing at 8 mg/kg IV once weekly (incl. one add. dose on Cycle 1 Day 4)
- 16 mg/kg QW: Dosing at 16 mg/kg IV once weekly (incl. one add. dose on Cycle 1 Day 4)
Arm/Group | 4 mg/kg QW | 8 mg/kg QW | 16 mg/kg QW
Number analyzed (Participants) | 4 | 14 | 39
µg/mL | 137.86 (79.43) | 311.67 (118.33) | 681.53 (226.69)

8. Secondary Outcome: Pharmacokinetics: AUC Cycle 1+2 - Area Under the Time/Concentration Curve for MOR202
Description: as for outcome 7
Time Frame: 56 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg*days/L
Arm/Group | 4 mg/kg QW | 8 mg/kg QW | 16 mg/kg QW
Number analyzed (Participants) | 4 | 14 | 39
mg*days/L | 3307.57 (2332.07) | 7970.15 (4289.21) | 18178.57 (8414.44)

ADVERSE EVENTS:
Time Frame: during the entire period of trial drug application and beyond until end of study visit/up to 30 days after last administration of study drug. Patients stayed on study drug up to 3 years.
Description: regular investigator assessment and laboratory testing
Groups:
- Part B: MOR03087 Weekly Dose Escalation: Treatment cycle 28 days, MOR03087 doses applied day 1, 8, 15 & 22 plus extra dose on day 4 of cycle 1, Initial MOR03087 dose 4 mg/kg, max 16 mg/kg For all parts, patients will be treated until PD or until a maximum of 3 years after first treatment.
  MOR03087: MOR03087 will be administered according to the Maximum Tolerated Dose (MTD) or recommended dose and dosing regimen for MOR03087 from parts A-E of the phase I dose escalation. The biweekly MOR03087 regimen as described in part A; the weekly regimen as described for parts B-E..
Arm/Group | Part A: MOR03087 Biweekly Dose Escalation | Part B: MOR03087 Weekly Dose Escalation | Part C: MOR03087 Plus Dexamethasone | Part D: MOR03087 Plus Pomalidomide + Dexamethasone | Part E: MOR03087 Plus Lenalidomide + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 2/31 | 0/4 | 0/18 | 1/21 | 4/17
Serious Adverse Events (participants affected / at risk) | 13/31 | 4/4 | 7/18 | 20/21 | 14/17
Other Adverse Events (participants affected / at risk) | 31/31 | 4/4 | 18/18 | 21/21 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: MOR03087 Biweekly Dose Escalation (N=31) | Part B: MOR03087 Weekly Dose Escalation (N=4) | Part C: MOR03087 Plus Dexamethasone (N=18) | Part D: MOR03087 Plus Pomalidomide + Dexamethasone (N=21) | Part E: MOR03087 Plus Lenalidomide + Dexamethasone (N=17)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 6 (9) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 3 (3) | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 (2) | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 1 (1)
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 1 (1)
Infusion-related reaction (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 0 | 1 (1) | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 | 0 | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 | 0 | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 (2) | 0 | 1 (2) | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 (3) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 | 0 | 1 (1) | 2 (2) | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 (0) | 0 | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 (0) | 0 | 1 (1)
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 (0) | 0 | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 0
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 | 0 | 0 | 0
Cardiovascular Disorder (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1)
Pericarditis (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 0
Cheast Pain (General disorders) | 0 | 0 | 0 | 0 | 1 (1)
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 (1)
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0
Infectious Pleural Effusion (Infections and infestations) | 0 | 0 (0) | 0 | 1 (1) | 0
Bacterial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Meningoencephalitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Parainfluenza Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Infection (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0
Respiratory Syncytal Virus Infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Varicella Zoster Virus Infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (2) | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1) | 0
Eccrine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (2) | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 (1)
Squamous Cell Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (2) | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: MOR03087 Biweekly Dose Escalation (N=31) | Part B: MOR03087 Weekly Dose Escalation (N=4) | Part C: MOR03087 Plus Dexamethasone (N=18) | Part D: MOR03087 Plus Pomalidomide + Dexamethasone (N=21) | Part E: MOR03087 Plus Lenalidomide + Dexamethasone (N=17)
Leukopenia (Blood and lymphatic system disorders) | 8 (13) | 4 (7) | 8 (28) | 17 (91) | 15 (55)
Nasopharyngitis (Infections and infestations) | 6 (8) | 1 (1) | 9 (12) | 4 (12) | 6 (10)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (12) | 8 (26) | 19 (113) | 12 (49)
Lymphopenia (Blood and lymphatic system disorders) | 5 (9) | 2 (4) | 8 (25) | 14 (43) | 13 (33)
Anaemia (Blood and lymphatic system disorders) | 13 (20) | 1 (3) | 7 (10) | 11 (34) | 6 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 6 (9) | 14 (51) | 11 (24)
C-reactive proteine increased (Investigations) | 0 (0) | 1 (2) | 3 (8) | 3 (10) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 4 (6)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (6)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 3 (14) | 0 (0) | 3 (3)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 2 (5) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Blood creatinine phosphokinase increased (Investigations) | 2 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 2 (10) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 6 (7) | 5 (10) | 6 (10)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (12) | 8 (18) | 4 (8)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 2 (2)
Bronchitis (Infections and infestations) | 4 (5) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (3) | 3 (3) | 2 (3) | 2 (3)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (3) | 3 (3) | 1 (1)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Fatigue (General disorders) | 11 (12) | 0 (0) | 6 (14) | 12 (22) | 6 (9)
Pyrexia (General disorders) | 5 (6) | 0 (0) | 3 (4) | 5 (7) | 2 (3)
Disease progression (General disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 3 (3)
Oedema peripheral (General disorders) | 3 (4) | 0 (0) | 2 (8) | 2 (3) | 4 (5)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (9) | 1 (1) | 4 (5) | 11 (15) | 10 (26)
Constipation (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 5 (8) | 11 (13)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 3 (4)
Nausea (Gastrointestinal disorders) | 10 (14) | 0 (0) | 2 (3) | 2 (10) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0) | 2 (7) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (5) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (16) | 2 (2) | 12 (12) | 9 (9) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 1 (1) | 2 (2) | 6 (11) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (7)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 2 (3) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (5) | 5 (9) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (7) | 7 (9) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (4) | 4 (6) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 4 (5) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 6 (8) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 3 (3) | 5 (8) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (8) | 0 (0) | 6 (8) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0) | 3 (5) | 1 (1) | 5 (6)
Paraesthesia (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 5 (13) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 3 (5) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 3 (9) | 5 (5) | 2 (4)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 3 (9) | 3 (6) | 3 (4)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 3 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 6 (21) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (3) | 3 (3) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Blood urea increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicous vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT01421186/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT01421186/SAP_001.pdf